CLINICAL TRIAL: NCT00235573
Title: Evaluation of Holotranscobalamin as an Indicator of Vitamin B12 Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 433-2005; 7591 (Other Grant/Funding Number: UF Clinical Research Center); M01RR000082 (NIH)
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Disorder of Vitamin B12
Keywords: Vitamin B12 absorption; Holo-transcobalamin
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin B12 supplement (Experimental): After taking a fasting blood sample, all subjects were given a light breakfast plus 9 micrograms of vitamin B12. Two more doses of vitamin B12 were administered 6 hours apart.
  Interventions: Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — After taking a fasting blood sample, all subjects were given a light breakfast plus 9 micrograms of vitamin B12. Two more doses of vitamin B12, 9 micrograms each, were administered 6 hours apart.

SUMMARY:
Vitamin B12 is an essential nutrient that the body needs for cells to divide and function normally. Individuals may develop a deficiency of vitamin B12 by either limiting the amount in the diet or by decreased vitamin B12 intake into the body (absorption). Keeping adequate B12 blood levels is important for health. Vitamin B12 deficiency may increase one's risk for developing anemia and can even lead to neurological problems and paralysis if the deficiency is severe and lasts a long time. It is very important for doctors to have accurate tests to determine if people are absorbing vitamin B12 normally so that treatment can be started before severe clinical problems occur.

The purpose of this research is to provide new information that may help scientists develop a better method to test for problems with absorbing vitamin B12. In this study, changes in the amounts of vitamin B12 bound to protein (transcobalamin) in the blood will be measured after doses of vitamin B12 are taken. If the amounts of this vitamin B12-protein complex (called holo-transcobalamin) change in response to taking a vitamin B12 supplement in normal individuals, it may be possible to use this information to develop a new sensitive test to identify individuals who have problems absorbing vitamin B12. This new vitamin B12 absorption test may be a better clinical test for vitamin B12 absorption than those now available for doctors to use.

DETAILED DESCRIPTION:
Part I Screening: Individuals who meet initial screening criteria will be scheduled to have fasting blood samples drawn in the General Clinical Research Center (GCRC). All participants will sign informed consent forms approved by the UF Institutional Review Board prior to the initiation of this part of the study. Subjects' heights and weights will be measured and subjects will be asked to complete a medical history questionnaire. Blood analyses will include serum B12, blood chemistry, and hematological indices. Females will be given a pregnancy test. Subjects eligible for Part II of the study (Intervention) will have serum B12 concentrations that are ≥444 pmol/L; will be non-anemic; and will have normal general blood chemistry (all values within or near the normal range), and no history of chronic disease (e.g., pernicious anemia, cancer, diabetes, renal disease, hypertension, neurological abnormalities, gastrointestinal disorders). Any subject with deficient (<148 pmol/L) serum B12 concentration [18] will not be eligible for participation and will be instructed to see their personal physician for complete follow-up and treatment.

Part II Intervention: Changes in B12 status assessment indicators in response to B12 supplementation will be evaluated.

Subjects will come to the GCRC the night before (Day 1) the intervention protocol. The next morning (Day 1) following an overnight fast, an indwelling catheter will be inserted from which repeated blood samples will be drawn throughout Day 1. A baseline fasting blood sample (#1) will be drawn. Subjects will then consume a light breakfast (including 1 piece of bread and 8 oz of orange juice) and will take a 9 ug dose of B12 (Dose 1). Thirty minutes after completion of the meal and consumption of the B12 supplement, a second blood sample (#2) will be drawn. Five subsequent hourly blood samples (# 3-7) will be drawn. After the 7th blood sample the subjects will consume one piece of bread and 8 ounces of orange juice and will take a second 9 ug dose of B12 (Dose 2) and have a blood sample (#8) drawn 30 minutes after consumption of the meal and the B12 dose. Five subsequent hourly blood samples (#9-13) will be drawn. The subjects will then consume one piece of bread and 8 ounces of orange juice and take a 9 ug dose of B12 (Dose 3). Another blood sample (#14) will be drawn 30 minutes after the meal and the B12 dose. One hour later, a final (Day 1) blood sample (#15) will be drawn followed by removal of the catheter. In addition to the bread and juice consumed with each B12 supplement, subjects will receive a mid-morning snack 2 hours after Dose 1 of the B12 supplement, lunch 3.5 hrs after Dose 1 of the B12 supplement, dinner at 4 hours after Dose 2 of the B12 supplement, and an evening snack at 3 hours after Dose 3. Low B12-containing foods will be provided in the GCRC. Water and non-caffeinated, non-caloric beverages will be allowed ad libitum.

The subjects will remain in the GCRC overnight and a fasting blood sample (#16) will be drawn in the morning on Day 2. On Day 2 participants will be provided breakfast following the blood draw, after which they will be free to leave the GCRC. Subjects will be provided with take-away meals and snacks (lunch, dinner, snacks) consisting of low-B12 containing foods.

Subjects will be instructed to return on the morning of Day 3 at which time they will have one am fasting blood sample (#17) drawn and will be provided with breakfast before they leave the GCRC. All overnight fasts will be from 10 pm the previous night. The following B12 indicators will be measured at each blood draw (a) holo-TC; (b) total-TC; (c) holo-HC and total HC; (d) serum B12; and (e) plasma albumin. Additional B12 status indicators (e.g. homocysteine, methylmalonic acid, RBC B12) will be measured at select blood draw intervals. A baseline folate analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* No vitamin B12-containing supplement use within past year
* No vitamin B12 injections within past year
* No use of tobacco products
* No chronic use of prescription medications except oral contraceptives
* No history of chronic disease (e.g., pernicious anemia, cancer, diabetes, renal disease, hypertension, neurological abnormalities, gastrointestinal disorders)
* BMI between 18.5-29.9
* General Chemistry Blood Tests (all values within or near normal range; hemoglobin if female ≥ 11.0 g/dL; if male ≥ 12 g/dL)
* B12 status (Serum B12 ≥ 444 pmol/L)
* Capable of understanding the informed consent form
* Agrees to comply with protocol requirements

Exclusion Criteria:

* History of pernicious anemia, cancer, diabetes, renal disease, hypertension, heart disease, neurological abnormalities, gastrointestinal disorders, lung disease, hepatic disease, hematologic, or other metabolic diseases that, in the opinion of the Co-Principal Investigators, would affect safety or compliance
* Vitamin B12 supplement use or injections within past year
* Pregnant or breast feeding
* Has BMI <18.5 or >29.9
* Has donated or lost a significant volume (>450 mL) of blood or plasma within 30 days of the study
* General chemistry lab values outside of ranges
* Serum B12 outside of range listed above
* Use of tobacco products
* Chronic use of prescription medications except oral contraceptives
* Does not understand the informed consent form
* Does not agree to comply with protocol requirements

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn B Bailey, PhD, Principal Investigator — University of Florida; Gail PA Kauwell, PhD, Principal Investigator — University of Florida
Locations (1):
- General Clinical Research Center, Shands Hospital, University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] von Castel-Dunwoody KM, Kauwell GP, Shelnutt KP, Vaughn JD, Griffin ER, Maneval DR, Theriaque DW, Bailey LB. Transcobalamin 776C->G polymorphism negatively affects vitamin B-12 metabolism. Am J Clin Nutr. 2005 Jun;81(6):1436-41. doi: 10.1093/ajcn/81.6.1436. PMID 15941899
- [Background] Bor MV, Nexo E, Hvas AM. Holo-transcobalamin concentration and transcobalamin saturation reflect recent vitamin B12 absorption better than does serum vitamin B12. Clin Chem. 2004 Jun;50(6):1043-9. doi: 10.1373/clinchem.2003.027458. Epub 2004 Mar 25. PMID 15044317
- [Background] Bor MV, Cetin M, Aytac S, Altay C, Nexo E. Nonradioactive vitamin B12 absorption test evaluated in controls and in patients with inherited malabsorption of vitamin B12. Clin Chem. 2005 Nov;51(11):2151-5. doi: 10.1373/clinchem.2005.055509. Epub 2005 Sep 15. PMID 16166166
- See also: The website for the UF General Clinical Research Center Clinical and Translational Science Institute — http://www.ctsi.ufl.edu/research/clinical-research-units/uf-clinical-research-center/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Gainesville/Alachua county area through newspaper ads, email, and flyers posted on the UF campus. Flyers also were given to individuals or groups. Respondents were interviewed by telephone and asked questions to ascertain if they met inclusion criteria. Individuals meeting criteria were screened for B12 status.
Pre-assignment Details: Individuals with a normal general blood chemistry profile, no history of chronic disease and normal CBC and vitamin B12 status were eligible to participate in the study. Those with deficient serum B12 levels were instructed to follow up with their personal physician. Subjects who met all inclusion criteria received the same treatment.
Groups:
- All Study Participants: All study participants received the same treatment of 3 doses of 9 micrograms of vitamin B12 at 6 hour intervals on day 1.
Period: Overall Study
Arm/Group | All Study Participants
Started | 21 (35 subjects screened; 14 not eligible; 21 started and completed study)
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Holo-transcobalamin
Description: Holo-TC is a vitamin B12 carrier protein. Only vitamin B12 bound to holo-TC can be taken up by cells. Changes in holo-TC after an oral dose of vitamin B12 may provide a clinical test to assess vitamin B12 absorption. The change in holo-transcobalamin (holo-TC) from baseline was measured at timed intervals in response to supplemental vitamin B12 and compared to baseline. The purpose was to ascertain the time point at which holo-TC reaches the maximum concentration in the blood following a dose of vitamin B12 in subjects without defects in vitamin B12 absorption.
Time Frame: Holo-transcobalamin measured at 24 hours after baseline
Population: The number of participants for analysis was per protocol.
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Vitamin B12 Group: All subjects received the same treatment of 3 doses of 9 micrograms of vitamin B12 at 6 hour intervals on day 1.
Arm/Group | Vitamin B12 Group
Number analyzed (Participants) | 21
pmol/L | 124 (46)

2. Secondary Outcome: Total Transcobalamin Measured at Intervals From Baseline to 48 Hours.
Time Frame: Baseline through 48 hours at intervals of 0, 0.5, 1.5, 2.5, 3.5, 4.5, 5.5, 6, 7, 8, 9, 10, 11, 11.5, 12.5, 24, 48
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pmol/L

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes